CLINICAL TRIAL: NCT05924425
Title: Daridorexant to Treat Insomnia in Patients With Mild Cognitive Impairment and Mild to Moderate Alzheimer Disease
Acronym: DARIDOR-ALZ
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RECHMPL22_0529
Record Dates: First submitted 2023-06-04; First posted 2023-06-29 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2023-06

CONDITIONS: Alzheimer Disease; Insomnia Disorder; Sleep
Keywords: Orexin; Daridorexant; Cognition; Alzheimer; Sleep; Insomnia
MeSH Terms: conditions — Alzheimer Disease; Sleep Initiation and Maintenance Disorders | interventions — daridorexant; Neuropsychological Tests

STUDY DESIGN:
Intervention Model Description: During Period A, patients randomized in the experimental group will receive the treatment every evening within 30 minutes of going to bed during one month. The treatment period will be followed by a one-week (range 5-12 days) washout period at home. During the second period (Period B), these patients will receive the placebo.
  During Period A, patients randomized in the control group will receive the placebo every evening within 30 minutes of going to bed during one month. The treatment period will be followed by a one-week (range 5-12 days) washout period at home. During the second period (Period B), these patients will receive the daridorexant 50 mg.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A randomization list will be generated and will remain confidential until the database is locked. Participants, investigators, and site personnel will be unaware of treatment allocation during the two crossover periods (Period A and Period B)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daridorexant 50 mg (Experimental): Patients will receive daridorexant 50 mg during one month (Period A or Period B).
  Daridorexant is an orally administered dual orexin type 1 and type 2 (OX1 and OX2) receptor antagonist (DORA) being developed for the treatment of insomnia.
  Interventions: Drug: Daridorexant 50 mg; Procedure: Polysomnography; Behavioral: Neuropsychological assessment; Behavioral: Questionnaires on sleep and behavioural problems; Procedure: Actimetrics; Procedure: 24-hour Ambulatory Blood Pressure Monitoring (ABPM; Other: Biomarker assay
- Placebo-controlled arm (Placebo Comparator): Patients will receive a placebo matching to daridorexant 50 mg during one month (Period A or Period B).
  Interventions: Drug: Placebo; Procedure: Polysomnography; Behavioral: Neuropsychological assessment; Behavioral: Questionnaires on sleep and behavioural problems; Procedure: Actimetrics; Procedure: 24-hour Ambulatory Blood Pressure Monitoring (ABPM; Other: Biomarker assay

INTERVENTIONS:
Drug: Daridorexant 50 mg — Patients randomized in the experimental group will receive the treatment every evening within 30 minutes of going to bed during one month. The treatment period (Period A or Period B) will be followed by a one-week (range 5-12 days) washout period at home.
  Arms: Daridorexant 50 mg
Drug: Placebo — Patients randomized in the control group will receive the placebo every evening within 30 minutes of going to bed during one month. The treatment period (Period A or Period B) will be followed by a one-week (range 5-12 days) washout period at home.
  Arms: Placebo-controlled arm
Procedure: Polysomnography — A full-night polysomnography recording with blood pressure and heart rate monitoring will be performed at night in the Sleep Laboratory from 11 p.m. to 7 a.m. at baseline (before the randomization) and at the end of each period (Period A/M1, Period B/M2). The recording procedure consists of an electroencephalogram, two electrooculograms, an electromyogram, an electrocardiogram, and a videographic recording. This examination is painless (the sensors are glued to the skin for the duration of the recording). The advantages of this video-polysomnography are based on the evaluation of sleep architecture, micro-arousals, respiratory events and nocturnal motor behavior.
Behavioral: Neuropsychological assessment — A full neuropsychological assessment will be performed at inclusion, M1, M2
Behavioral: Questionnaires on sleep and behavioural problems — Questionnaires on sleep and behavioural problems will be performed at inclusion, M1, M2
Procedure: Actimetrics — Measurement of actimetrics for seven days in average (with a minimum of three nights required) prior to the inclusion visit, M1 visit and M2 visit.
Procedure: 24-hour Ambulatory Blood Pressure Monitoring (ABPM — Evaluation of the 24-hour hemodynamic profile of a patient by multiple and regular blood pressure and heart rate measurements. The ABP will be monitored at inclusion, M1 and M2
Other: Biomarker assay — Determination of AD biomarkers (Aβ42, Aβ40, Tau, P-Tau, neurofilament) and proinflammatory cytokines (TNFa, IL6) in serum and cerebrospinal fluid (CSF) and dosage of Orexin-A/hypocretin-1 in the CSF

SUMMARY:
DARIDOR-ALZ is a phase IV clinical trial designed to evaluate both the efficacy and safety of daridorexant, a selective dual orexin receptor antagonist that blocks the actions of the orexin neuropeptides at both orexin-1 and orexin-2 receptors, in selected populations of MCI and mild-to-moderate AD patients with insomnia complaints.

DETAILED DESCRIPTION:
This Phase IV clinical trial is a monocentric, randomized, double-blind, placebo-controlled, 2 way-crossover study (with two periods of one month separated by a washout period range from 5 to 12 days).The study population includes MCI and mild-to-moderate AD patients aged between 60 and 85 years old, with insomnia complaints.

A single-night baseline polysomnography recording will be performed from 11 pm to 7 am at the Montpellier Sleep Unit. After a baseline PSG that assessed TST < 6 hours and WASO > 1 hour, treatment will be assigned using an interactive response technology system.

A randomization list will be generated and will remain confidential until the database is locked. Participants, investigators, and site personnel will be unaware of treatment allocation during the two crossover periods. Patients will be randomized (1:1) to receive daridorexant 50 mg or placebo, without titration, every evening within 30 minutes of going to bed during both treatment periods (Treatment Period A and B) of one-month duration each. Each treatment period will be followed by a one-week (range 5-12 days) washout period at home.

A ten-month open-label (OL) study with daridorexant 50 mg will be proposed to all participants after completing the second treatment period. Based on the experience with another DORA study in patients with mild-to-moderate probable Alzheimer's disease, the investigators would need to recruit 62 patients (including drop-outs).

ELIGIBILITY:
Inclusion criteria :

* Age [60-85] years old
* Outpatients
* Pre-screening:

  * Complaints of dissatisfaction with sleep quantity or quality, despite adequate opportunity for sleep, at least 3 nights per week and for at least 3 months, and
  * Total sleep time causes clinically significant distress or impairment in daytime functioning, and
  * Total sleep time estimated by interview and sleep diary was below 6 hours, on at least 3 nights per week and for at least 1 month before screening, and
  * Insomnia Severity Scale ISI© score ≥ 15
* Baseline PSG (at randomization) assessed TST < 6 hours and WASO > 1 hour
* Diagnosis of MCI and AD patients at an early stage according to the NIA diagnosis criteria (core clinical criteria for MCI, positive biomarker for CSF Aβ42 and neuronal injury (hippocampal and/or temporal atrophy by MRI))
* MMSE from 12 to 26
* Clinical Dementia Rating CDR from 0.5 to 2
* Possible of CNS drugs if stable dose for at least 3 months: anticholinesterase drugs (rivastigmine, donepezil, galantamine) or memantine
* For a male subject who is not sterilized and is sexually active with a female partner of childbearing potential, no contraceptive methods are needed

Non inclusion criteria :

* Patients significantly dependent on caregivers
* Institutionalized patients
* Analphabetism or subjects unable to read or/and write
* Patients unable to perform the neuropsychological tests
* Patients unable to complete the study instruments (sleep diary)
* Planned longer stay outside the region that prevents compliance with the visit schedule
* Patients who cannot be followed up for at least 2 months
* History of narcolepsy and/or cataplexy
* History of drug or alcohol abuse or addiction
* History of depression or suicidal ideation/attempt or other psychiatric conditions
* Moderate and severe liver failure
* PSG baseline evidence of significant/severe sleep-related breathing disorder (defined as >30 apnea/hypopnea episodes per hour)
* Treatments interfering with sleep-wake patterns
* Psychotropic drugs: antidepressants (SSRI (e.g. fluoxetine, sertraline, paroxetine…), SNRI (e.g. venlafaxine, duloxetine)), neuroleptics (e.g. clozapine, olanzapine, aripiprazole...), and hypnotics (benzodiazepines, zolpidem, zopiclone) or drug for pain (level 2 (e.g. codeine, tramadol), and level 3 (morphine and derivatives))
* Hypersensitivity to the active substance or to any of the excipients listed in the Summary of Product Characteristics (SmPC)
* Forbidden and restricted concomitant medications:

  * Concomitant CNS-depressant medicinal products
  * CYP3A4 inhibitors
  * CYP3A4 inducers
* Participation in another clinical trial or administration of an investigational product
* Protected population according to articles of the French Public Health Code (e.g. patients under law protection, prisoners, pregnant, parturient or lactating women, and patients under guardianship/curatorship).
* Subjects not covered by public health insurance
* Failure to obtain written informed consent after a reflection period

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2026-05-13 (Estimated); Study Completion 2027-03-13 (Estimated)

PRIMARY OUTCOMES:
Change in Total Sleep Time (TST). | from baseline to the end of each period A/B (Month1/Month2)
  TST is defined as the total sleep time in minutes. The total sleep time is the total amount of sleep time scored during the total recording time. The TST is measured during polysomnography.

SECONDARY OUTCOMES:
Change in the wake time after sleep onset (WASO) | from baseline to the end of each period A/B (Month1/Month2)
  WASO is defined as the time to wake after initial sleep onset. WASO is measured during overnight sleep laboratory (PSG) assessment and defined as the duration of wakefulness from the onset of persistent sleep.
Change in Latency to Persistent Sleep (LPS) | from baseline to the end of each period A/B (Month1/Month2)
  LPS is the time in minutes from 'lights out' that marks the starting of total recording time to the first epoch recorded as sleep. The LPS is measured during polysomnography.
Measure of sleep time at stage 1-2 during polysomnography | from baseline to the end of each period A/B (Month1/Month2)
  Time spent in stage 1-2 sleep measured in hours and minutes during polysomnography.
Measure of sleep time at stage 3 during polysomnography | from baseline to the end of each period A/B (Month1/Month2)
  Time spent in stage 3 sleep measured in hours and minutes during polysomnography.
Measure of number of wake bouts on the whole night | from baseline to the end of each period A/B (Month1/Month2)
  The number of wake bouts on the whole night will be measured by polysomnography.
Measure of number of wake bouts per quarter of the night | from baseline to the end of each period A/B (Month1/Month2)
  The number of wake bouts per quarter of the night will be measured by polysomnography.
Changes in sleep and wake duration | from baseline to the end of each period A/B (Month1/Month2)
  Average sleep duration (in hours and minutes) over a 7-day period from inclusion to each visit measured by actimetry.
Changes in sleep and wake duration | from baseline to Month 6
  Average sleep duration (in hours and minutes) over a 7-day period from inclusion to each visit measured by actimetry.
Changes in sleep and wake duration | from baseline to Month 12
  Average sleep duration (in hours and minutes) over a 7-day period from inclusion to each visit measured by actimetry.
Variations in the results of self-reported questionnaires administered to patients - Insomnia Severity Index (ISI) | from baseline to the end of each period A/B (Month1/Month2)
  Values and variations from baseline of patient-reported outcomes including self-reported questionnaire ISI.
  The Insomnia Severity Index (ISI) is a 7-item self-report questionnaire assessing the nature, severity of both nighttime and daytime components of insomnia, and impact of insomnia.
  Each item is scored 0 (no problem) - 4 (very big problem) with total between 0-28 (absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Variations in the results of self-reported questionnaires administered to patients - Insomnia Severity Index (ISI) | from baseline to Month 6
  Values and variations from baseline of patient-reported outcomes including self-reported questionnaire ISI.
  The Insomnia Severity Index (ISI) is a 7-item self-report questionnaire assessing the nature, severity of both nighttime and daytime components of insomnia, and impact of insomnia.
  Each item is scored 0 (no problem) - 4 (very big problem) with total between 0-28 (absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Variations in the results of self-reported questionnaires administered to patients - Insomnia Severity Index (ISI) | from baseline to Month 12
  Values and variations from baseline of patient-reported outcomes including self-reported questionnaire ISI.
  The Insomnia Severity Index (ISI) is a 7-item self-report questionnaire assessing the nature, severity of both nighttime and daytime components of insomnia, and impact of insomnia.
  Each item is scored 0 (no problem) - 4 (very big problem) with total between 0-28 (absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Variations in the results of self-reported questionnaires administered to patients - Epworth Sleepiness Scale (ESS) | from baseline to the end of each period A/B (Month1/Month2)
  Values and variations from baseline of patient-reported outcomes including self-reported questionnaire ESS.
  The Epworth Sleepiness Scale (ESS) is a self-report measure of daytime sleepiness in various situations and consists of eight questions. ESS score can range from 0 to 24 (1 to 6 points: Normal sleep; 7 to 8 points: Average sleepiness: 9 to 24 points: Abnormal (possibly pathologic) sleepiness).
Variations in the results of self-reported questionnaires administered to patients - ESS | from baseline to Month 6
  Values and variations from baseline of patient-reported outcomes including self-reported questionnaire ESS.
  The Epworth Sleepiness Scale (ESS) is a self-report measure of daytime sleepiness in various situations and consists of eight questions. ESS score can range from 0 to 24 (1 to 6 points: Normal sleep; 7 to 8 points: Average sleepiness: 9 to 24 points: Abnormal (possibly pathologic) sleepiness).
Variations in the results of self-reported questionnaires administered to patients - Epworth Sleepiness Scale (ESS) | from baseline to Month 12
  Values and variations from baseline of patient-reported outcomes including self-reported questionnaire ESS.
  The Epworth Sleepiness Scale (ESS) is a self-report measure of daytime sleepiness in various situations and consists of eight questions. ESS score can range from 0 to 24 (1 to 6 points: Normal sleep; 7 to 8 points: Average sleepiness: 9 to 24 points: Abnormal (possibly pathologic) sleepiness).
Variations in the results of self-reported questionnaires administered to patients - Insomnia Daytime Symptoms and Impacts (IDSIQ) | from baseline to the end of each period A/B (Month1/Month2)
  Values and variations from baseline of patient-reported outcomes including self-reported questionnaire IDSIQ.
  The Insomnia Daytime Symptoms and Impacts Questionnaire (IDSIQ) is a patient-reported outcome instrument that assesses daytime functioning in patients with insomnia.
  It consists of 14 items (each using a numeric rating scale from 0 to 10) grouped into 3 domains : Alert/Cognition, Mood, and Sleepiness domain reflecting daytime impairment of insomnia.
  The IDSIQ sleepiness domain has 4 items, and the domain score ranges from 0 to a maximum of 40, where a higher score indicates a greater burden. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Variations in the results of self-reported questionnaires administered to patients - Insomnia Daytime Symptoms and Impacts (IDSIQ) | from baseline to Month 6
  Values and variations from baseline of patient-reported outcomes including self-reported questionnaire IDSIQ.
  The Insomnia Daytime Symptoms and Impacts Questionnaire (IDSIQ) is a patient-reported outcome instrument that assesses daytime functioning in patients with insomnia.
  It consists of 14 items (each using a numeric rating scale from 0 to 10) grouped into 3 domains : Alert/Cognition, Mood, and Sleepiness domain reflecting daytime impairment of insomnia.
  The IDSIQ sleepiness domain has 4 items, and the domain score ranges from 0 to a maximum of 40, where a higher score indicates a greater burden. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Variations in the results of self-reported questionnaires administered to patients - Insomnia Daytime Symptoms and Impacts (IDSIQ) | from baseline to Month 12
  Values and variations from baseline of patient-reported outcomes including self-reported questionnaire IDSIQ.
  The Insomnia Daytime Symptoms and Impacts Questionnaire (IDSIQ) is a patient-reported outcome instrument that assesses daytime functioning in patients with insomnia.
  It consists of 14 items (each using a numeric rating scale from 0 to 10) grouped into 3 domains : Alert/Cognition, Mood, and Sleepiness domain reflecting daytime impairment of insomnia.
  The IDSIQ sleepiness domain has 4 items, and the domain score ranges from 0 to a maximum of 40, where a higher score indicates a greater burden. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Variations in the results of self-reported questionnaires administered to patients - Sleep Diaries | from baseline to the end of each period A/B (Month1/Month2)
  Values and variations from baseline of patient-reported outcomes including self-reported questionnaire Sleep diaries.
  Participants will completed a daily sleep diary (sleep onset latency, wake after sleep onset, early morning awakening, total wake time, total sleep time, and sleep efficiency).
Variations in the results of self-reported questionnaires administered to patients - Sleep Diaries | from baseline to Month 6
  Values and variations from baseline of patient-reported outcomes including self-reported questionnaire Sleep diaries.
  Participants will completed a daily sleep diary (sleep onset latency, wake after sleep onset, early morning awakening, total wake time, total sleep time, and sleep efficiency).
Variations in the results of self-reported questionnaires administered to patients - Sleep Diaries | from baseline to Month 12
  Values and variations from baseline of patient-reported outcomes including self-reported questionnaire Sleep diaries.
  Participants will completed a daily sleep diary (sleep onset latency, wake after sleep onset, early morning awakening, total wake time, total sleep time, and sleep efficiency).
Variations in the results of health assessment questionnaires administered to patients - Neuropsychiatric Inventory (NPI) | from baseline to the end of each period A/B (Month1/Month2)
  The nocturnal agitation will be assessed by using the Neuropsychiatric Inventory (NPI) agitation/aggression domain.
  The Neuropsychiatric Inventory (NPI), which consists of 12 items scored with questions, sub-questions, and frequency and severity ratings, is used to assess behavioral changes in Alzheimer disease and other neurodegenerative disorders. The agitation/aggression domain will be evaluated at each visit.
Variations in the results of health assessment questionnaires administered to patients - Neuropsychiatric Inventory (NPI) | from baseline to Month 6
  The nocturnal agitation will be assessed by using the Neuropsychiatric Inventory (NPI) agitation/aggression domain.
  The Neuropsychiatric Inventory (NPI), which consists of 12 items scored with questions, sub-questions, and frequency and severity ratings, is used to assess behavioral changes in Alzheimer disease and other neurodegenerative disorders. The agitation/aggression domain will be evaluated at each visit.
Variations in the results of health assessment questionnaires administered to patients - Neuropsychiatric Inventory (NPI) | from baseline to Month 12
  The nocturnal agitation will be assessed by using the Neuropsychiatric Inventory (NPI) agitation/aggression domain.
  The Neuropsychiatric Inventory (NPI), which consists of 12 items scored with questions, sub-questions, and frequency and severity ratings, is used to assess behavioral changes in Alzheimer disease and other neurodegenerative disorders. The agitation/aggression domain will be evaluated at each visit.
Variations in the results of health assessment questionnaires administered to patients - Beck Depression Inventory (BDI) | from baseline to the end of each period A/B (Month1/Month2)
  Values and variations from baseline of patient-reported outcomes including health assessment questionnaire BDI.
  The Beck Depression Inventory (BDI) contains 21 items on a 4-point scale from 0 (symptom absent) to 3 (severe symptoms). The minimum score is 0 and the maximum score is 63, with a higher score indicating more severe depressive symptoms.
Variations in the results of health assessment questionnaires administered to patients - Beck Depression Inventory (BDI) | from baseline to Month 6
  Values and variations from baseline of patient-reported outcomes including health assessment questionnaire BDI.
  The Beck Depression Inventory (BDI) contains 21 items on a 4-point scale from 0 (symptom absent) to 3 (severe symptoms). The minimum score is 0 and the maximum score is 63, with a higher score indicating more severe depressive symptoms.
Variations in the results of health assessment questionnaires administered to patients - Beck Depression Inventory (BDI) | from baseline to Month 12
  Values and variations from baseline of patient-reported outcomes including health assessment questionnaire BDI.
  The Beck Depression Inventory (BDI) contains 21 items on a 4-point scale from 0 (symptom absent) to 3 (severe symptoms). The minimum score is 0 and the maximum score is 63, with a higher score indicating more severe depressive symptoms.
Variations in the results of health assessment questionnaires administered to patients - EuroQoL-5D (EQ5D) | from baseline to the end of each period A/B (Month1/Month2)
  Values and variations from baseline of patient-reported outcomes including health assessment questionnaire EQ5D.
  The EuroQol 5-dimensional descriptive system (EQ5D) is a Health Assessment Scale quality of life questionnaire evaluating: mobility, washing and dressing, daily activities, pain and anxiety. Each question has 3 levels of answers: No problem, some problems and important problems. Lower score indicate better outcomes.
  The questionnaire also includes a visual analog scale in which the patient quantifies his or her perception of quality of life using a score ranging from the worst imaginable state of health (0) to the best imaginable state of health (100).
Variations in the results of health assessment questionnaires administered to patients - EuroQoL-5D (EQ5D) | from baseline to Month 6
  Values and variations from baseline of patient-reported outcomes including health assessment questionnaire EQ5D.
  The EuroQol 5-dimensional descriptive system (EQ5D) is a Health Assessment Scale quality of life questionnaire evaluating: mobility, washing and dressing, daily activities, pain and anxiety. Each question has 3 levels of answers: No problem, some problems and important problems. Lower score indicate better outcomes.
  The questionnaire also includes a visual analog scale in which the patient quantifies his or her perception of quality of life using a score ranging from the worst imaginable state of health (0) to the best imaginable state of health (100).
Variations in the results of health assessment questionnaires administered to patients - EuroQoL-5D (EQ5D) | from baseline to Month 12
  Values and variations from baseline of patient-reported outcomes including health assessment questionnaire EQ5D.
  The EuroQol 5-dimensional descriptive system (EQ5D) is a Health Assessment Scale quality of life questionnaire evaluating: mobility, washing and dressing, daily activities, pain and anxiety. Each question has 3 levels of answers: No problem, some problems and important problems. Lower score indicate better outcomes.
  The questionnaire also includes a visual analog scale in which the patient quantifies his or her perception of quality of life using a score ranging from the worst imaginable state of health (0) to the best imaginable state of health (100).
Change in cognition | from baseline to the end of each period A/B (Month1/Month2)
  The Alzheimer's Disease Cooperative Study - Preclinical Alzheimer Cognitive (ADCS-PACC) scale score will be based on scores from the Mini Mental State Examination (MMSE) (range from 0-30 points), Free and Cued Selective Reminding Test - FCSRT (range from 0-48 points), the Digit Substitution Symbol Test, the Wechsler Intelligence Scale for Adults (WAIS-IV) (range from 0-93 points), the Clinical Dementia Rating Scale (CDR) (range from 0-18 points), and the 2-minute Verbal Fluency Test.
  The ADCS-PACC will be measured at each visit. Each of the component change scores is divided by the baseline sample standard deviation of that component, to form standardized z scores. These z scores are summed to form the composite. Z Scores could range from -5 to +5 with higher scores indicating less deficit and lower scores indicating greater deficit.
Change in cognition | from baseline to Month 6
  The Alzheimer's Disease Cooperative Study - Preclinical Alzheimer Cognitive (ADCS-PACC) scale score will be based on scores from the Mini Mental State Examination (MMSE) (range from 0-30 points), Free and Cued Selective Reminding Test - FCSRT (range from 0-48 points), the Digit Substitution Symbol Test, the Wechsler Intelligence Scale for Adults (WAIS-IV) (range from 0-93 points), the Clinical Dementia Rating Scale (CDR) (range from 0-18 points), and the 2-minute Verbal Fluency Test.
  The ADCS-PACC will be measured at each visit. Each of the component change scores is divided by the baseline sample standard deviation of that component, to form standardized z scores. These z scores are summed to form the composite. Z Scores could range from -5 to +5 with higher scores indicating less deficit and lower scores indicating greater deficit.
Change in cognition | from baseline to Month 12
  The Alzheimer's Disease Cooperative Study - Preclinical Alzheimer Cognitive (ADCS-PACC) scale score will be based on scores from the Mini Mental State Examination (MMSE) (range from 0-30 points), Free and Cued Selective Reminding Test - FCSRT (range from 0-48 points), the Digit Substitution Symbol Test, the Wechsler Intelligence Scale for Adults (WAIS-IV) (range from 0-93 points), the Clinical Dementia Rating Scale (CDR) (range from 0-18 points), and the 2-minute Verbal Fluency Test.
  The ADCS-PACC will be measured at each visit. Each of the component change scores is divided by the baseline sample standard deviation of that component, to form standardized z scores. These z scores are summed to form the composite. Z Scores could range from -5 to +5 with higher scores indicating less deficit and lower scores indicating greater deficit.
Change in blood pressure | from baseline to the end of each period A/B (Month1/Month2)
  Decrease in blood pressure variability (Systolic and Diastolic) during polysomnography and increase in 24-hour blood pressure monitoring dipping pattern from baseline to the end of each period (Month 1/Month 2) comparing daridorexant 50 mg with placebo.
Change in blood pressure | from baseline to Month 6
  Change in 24-hour blood pressure (Systolic and Diastolic) monitoring dipping pattern from baseline to the month 6 with daridorexant 50 mg.
Change in blood pressure | from baseline to Month 12
  Change in 24-hour blood pressure (Systolic and Diastolic) monitoring dipping pattern from baseline to the month 12 with daridorexant 50 mg.
Change in blood AD biomarkers and proinflammatory cytokines levels | from baseline to the end of each period A/B (Month1/Month2)
  Determination of blood AD biomarkers (Aβ42, Aβ40, Tau, P-Tau, neurofilament) and proinflammatory cytokines (TNFa, IL6) levels in serum.
Change in blood AD biomarkers and proinflammatory cytokines levels | from baseline to Month 6
  Determination of blood AD biomarkers (Aβ42, Aβ40, Tau, P-Tau, neurofilament) and proinflammatory cytokines (TNFa, IL6) levels in serum.
Change in blood AD biomarkers and proinflammatory cytokines levels | from baseline to Month 12
  Determination of blood AD biomarkers (Aβ42, Aβ40, Tau, P-Tau, neurofilament) and proinflammatory cytokines (TNFa, IL6) levels in serum.
Concentration of CSF AD biomarkers and proinflammatory cytokines | baseline
  Determination of AD biomarkers (Aβ42, Aβ40, Tau, P-Tau, neurofilament) and proinflammatory cytokines (TNFa, IL6) levels in cerebrospinal fluid (CSF).
Concentration of CSF orexinA/hypocretin | baseline
  Determination orexinA/hypocretin in cerebrospinal fluid (CSF)
Percentage of Serious Adverse Events Occurring | between baseline and 12 months
  Safety: rates of serious adverse events between baseline and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Dauvilliers, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital, Montpellier, Montpellier, France